CLINICAL TRIAL: NCT03350776
Title: Pilot Observational and Analytic Study of Practices and Organizations Related to Emerging Occupations of Care Coordination in Oncology: Modeling the Concept of Care Coordination in Oncology (EPOCK)
Brief Title: Practices and Organizations Related to Emerging Occupations of Care (EPOCK) Coordination in Oncology
Acronym: EPOCK
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2016/31
Record Dates: First submitted 2017-11-09; First posted 2017-11-22 (Actual); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Care Coordination in Oncology
Keywords: Neoplasm; Chronic disease; Complex cases; Care coordination; Oncologic nursing; Theoretical model
MeSH Terms: conditions — Neoplasms; Chronic Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Care coordination — Care coordination and associated emerging occupations by comparing theoretical expected outcomes to professionals, patients and caregivers representations

SUMMARY:
Several stakeholders are implied in cancer care pathways and there is a need for coordinating their actions. New occupations of care coordination have thus emerged. However, the conditions of their efficiency have been too few reported and included discrepancies between reports. In this context, the main objective is to propose a modeling of care coordination and associated emerging occupations (nurse-based) by comparing theoretical expected outcomes to professionals, patients and caregivers representations.

DETAILED DESCRIPTION:
Several stakeholders are implied in cancer care pathways and there is a need to coordinate their actions. New occupations of care coordination have thus emerged, such as nurse coordinator in France (IDEC: Infirmière de Coordination). However, the conditions of their efficiency are not well known. Moreover, several other complementary approaches and nurse occupations have to be identified because of their contribution to care coordination (IDE TAS, IPO, IDE AMA, IDE-CO, IDE HAD-CAD, IDE ETP)*. Finally, all together, these interventions of care coordination appeared as complex and asked for a theoretical model. Because of this high variability of the practices, without an underlying model, the impact of care coordination on patient quality of life, safety and efficiency of care is difficult to assess. In this context, the main objective is to propose a modeling of care coordination and associated emerging occupations by comparing theoretical expected outcomes to professionals, patients and caregivers representations.

The pilot observational study is based on three distinct stages: (1) the definition of care coordination in oncology using a literature review and a Delphi consensus study; (2) the description of practices, contexts, perceptions and attitudes related to care coordination occupations in oncology using a qualitative and a cross-sectional quantitative survey; (3) the comparison of the practices to the theoretical model to propose a modeling of care coordination occupations in oncology.

ELIGIBILITY:
Inclusion Criteria:

* For health institutions: public or private institutions in which nurses contributing to care coordination. Each institution will be associated with one type of coordination occupation, even if other healthcare workers contribute to care coordination in the same institution.
* For professionals of care coordination: nurses contributing to care coordination in oncology (IDEC , IDE TAS, IPO, IDE AMA, IDE-CO, IDE HAD-CAD or IDE ETP)
* For professionals working with professionals of care coordination:

  * Medical and non-medical healthcare professionals (oncologist, surgeon, nurses…), administrative professionals (secretary…), professionals of supportive care (psychologists, social workers…) and volunteers in patient organizations.
  * Private practitioners: general practitioner, private nurses, pharmacist
* For the patients : adults under supervision of the selected professionals of care coordination for at least four weeks and able to express themselves
* For the caregivers: family caregivers of the selected patients.

Exclusion Criteria:

* For health institutions: private healthcare networks, territorial support platforms, home-based care providers, healthcare houses
* For professionals of care coordination: coordinating medical doctors of care networks, coordinating medical doctors of hospital care at home, practitioners of regional cancer networks.
* For the patients: <18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Four samples :
  * Professionals of cancer care coordination
  * Cancer patients
  * Family caregivers of the selected patients
  * Professionals working with professionals of care coordination
Sampling Method: Non-Probability Sample
Enrollment: 960 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2019-10-02 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Modeling of care coordination in Oncology in France | During the whole period (36 months: from Month 1 to Month 36)
  Constitutive elements of modelling of care coordination in oncology in France (qualitative analysis)

SECONDARY OUTCOMES:
Care coordination profesionals quality of life | Quantitative cross sectional survey (from Month 10 to Month 29)
  Three scores : perceived organizational support, role conflict and commitment to the organization
Satisfaction with care coordination for profes professionals working with professionals of care coordination | Quantitative cross sectional survey (from Month 10 to Month 29)
  Score of satisfaction
Patients quality of life and satisfaction with care coordination | Quantitative cross sectional survey (from Month 10 to Month 29)
  Score of satisfaction and score of quality of life (measured with the European Organization for Research and Treatment (EORTC) quality of life questionnaire)
Caregivers burden with care coordination | Quantitative cross sectional survey (from Month 10 to Month 29)
  Score of burdean (Zarit Burden Interview) with care coordination
Caregivers satisfaction with care coordination | Quantitative cross sectional survey (from Month 10 to Month 29)
  Score of satisfaction with care coordination

CONTACTS AND LOCATIONS:
Locations (10):
- France (10):
  - Institut Sainte Catherine, Avignon
  - CHU de Bordeaux, Bordeaux
  - Clinique Tiivoli Ducos, Bordeaux
  - CH Sud Gironde, Langon
  - CH de Libourne, Libourne
  - Institut Curie, Paris
  - Institut de Cancérologie de la Loire, Saint-Priest
  - HAD Bagatelle, Talence
  - CHU de Toulouse, Toulouse
  - Institut Claudius Regaud, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Colombani F, Calcagni N, Sibe M, Kret M, Fournier H, Ravaud A, Quintard B, Saillour-Glenisson F. Evidence-based modelling and taxonomy of hospital-based cancer care coordination nurses' roles and boundaries: an iterative multiphase convergent mixed study. BMJ Oncol. 2025 Nov 18;4(1):e000771. doi: 10.1136/bmjonc-2025-000771. eCollection 2025. PMID 41323425
- [Derived] Colombani F, Sibe M, Kret M, Quintard B, Ravaud A, Saillour-Glenisson F. EPOCK study protocol: a mixed-methods research program evaluating cancer care coordination nursing occupations in France as a complex intervention. BMC Health Serv Res. 2019 Jul 12;19(1):483. doi: 10.1186/s12913-019-4307-7. PMID 31299966